CLINICAL TRIAL: NCT05830331
Title: Enhanced Recovery After Spine Surgery (ERASS) Versus Traditional Spine Surgical Care (TC): A Randomized, Prospective Trial
Brief Title: Enhanced Recovery After Spine Surgery Randomized Clinical Trial
Acronym: ERASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Zarina Ali, Chief, Penn Presbyterian Medical Center Department of Neurosurgery, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 831303
Record Dates: First submitted 2023-03-01; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: ERAS

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Treatment (Experimental)
  Interventions: Other: ERASS Pathway

INTERVENTIONS:
Other: ERASS Pathway — Enhanced Recovery After Spinal Surgery
  Arms: Treatment

SUMMARY:
The purpose of this study is to compare two different approaches to the care patients receive before, during and after their spinal surgery and to determine if either approach has a significant difference in patient outcomes, opioid use, and recovery following spine surgery. The study will compare the standard-of-care surgical approach taken at the Hospital of the University of Pennsylvania with the Enhanced Recovery After Spine Surgery (ERASS) pathway. ERASS is a program that will provide additional education before your surgery, reduce your opioid consumption, and provide earlier physical therapy than you would normally receive under the standard-of-care approach, among other protocols outlined in this consent. Patients will be randomized to receive either of these approaches and the researchers will collect information to better understand if the ERASS approach provides more patient benefits.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 and older (both male and female), who present to the department of neurosurgery at the Hospital of the University of Pennsylvania and who are determined to require elective spine surgery with one of two senior spine neurosurgeons, Drs. Malhotra and Marcotte.

Exclusion Criteria:

* Patients who are pregnant
* Incarceration
* Patients under the age of 18
* Patients unable to participate in the consent procedure
* Patients undergoing emergent surgery
* Patients with liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2021-10-13 (Actual)

PRIMARY OUTCOMES:
Opioid use during hospitalization | post-operative days during hospital admission, up to 20 days
  Total opioid use during hospitalization after surgery
Opioid use after surgery | up to one month after surgery
  Proportion of patients using opioids one month after surgery

SECONDARY OUTCOMES:
Total Opioid Consumption During Hospitalization Using Morphine Equivalents | post-operative days during hospital admission, up to 20 days
  * Total morphine equivalents for each post-operative day (POD) 0, 1, 2, 3...21+
  * Total morphine equivalents for all post-operative days
Usage of PCA during hospitalization | from admission to discharge, up to 20 days
  • Patient-controlled analgesia (PCA) use (collected mg per hour and morphine equivalent)
Opioid Consumption During Hospitalization | post-operative days during hospital admission, up to 20 days
  * Use of intravenous (IV) narcotics (collected by "Yes" or "No")
  * Use of Narcan/Naloxon (collected by "Yes" or "No")
Opioid Refills After Surgery | up to one month after surgery
  • Number of times opioid was refilled over 1 month
Opioid Prescribed After Surgery | up to one month after surgery
  • Medications and number of pills prescribed at discharge
Opioid Refills (days) After Surgery | up to one month after surgery
  • Number of days until 1st, 2nd, and 3rd refill
Opioids Left Over After Surgery | up to one month after surgery
  • Number of pills leftover at one-month timepoint from surgery
Opioid Compliance During Hospitalization | from admission to discharge, up to 20 days
  • Compliance with inpatient Enhanced Recovery After Surgery (ERAS) multimodal pain regimen
Pain Control Medication Usage | post-operative days during hospital admission, up to 20 days
  Total usage of non-opioids medication was collected by mg with the following medications:
  * Acetaminophen
  * Dexamethasone
  * Lidocaine/ Lidoderm
  * Toradol
  * Valium
  * Flexeril
  * Gabapentin
  * Pregabalin
  * Ketamine
Pain Control Measurement | from admission to discharge, up to 20 days
  Using the Visual Analogue Scale (VAS), patients had to rate their pain on a scale of 1 to 10, with 1 being the least pain and 10 being the least amount of pain. Timepoints included:
  * Preop pain score
  * Discharge pain score
  * Average pain score
  * Minimum pain score
  * Maximum pain score
Mobilization During Hospitalization | post-operative days 0 and 1 during hospital admission
  * Collection of patient mobilization post-operative day (POD) 0, 1
  * Collection of patient ambulation post-operative day (POD) 0, 1
Time to Mobilization During Hospitalization | post-operative days during hospital admission, up to 20 days
  • Record time to mobilization and ambulation
Patient Falls | from admission to discharge, up to 20 days
  • Collection of total number of inpatient falls
Usage of Foley During Hospitalization Course | from admission to discharge, up to 20 days
  • Collection of patient use of Foley catheter post-operatively
Usage of Straight Catheterization During Hospitalization Course | from admission to discharge, up to 20 days
  • Collection of patient use for straight catheterization post-operatively
Collection of Inpatient Status | from admission to discharge, up to 20 days
  • Collection of patient hospitalization status post-operatively including: inpatient, outpatient and observational
Length of Stay (days) | from admission to discharge, up to 20 days
  * Total length of stay (days) in hospital
  * Total length of stay (days) in intensive care unit (ICU)
Length of Stay (hours) | from admission to discharge, up to 20 days
  * Total length of stay (hours) in hospital
  * Total length of stay (hours) in intensive care unit (ICU)
Collection of Patient Complications | from admission to discharge, up to 20 days and up to 6 months after surgery
  Collection of complications (Yes/No) including:
  * Death
  * Complications (including surgical site infection, urinary tract infections, cardiopulmonary events, wound dehiscence rates, and non-union rates, and others)
  * Morbidities
Collection of Patient Re-admissions After Discharge | up to 3 months after surgery
  * Collection of patient re-admission 30-days after surgery
  * Collection of patient re-admission 90-days after surgery
Collection of Re-operation After Surgery | up to 3 months after surgery
  • Collection of any reoperations that occurred after the patient's initial surgery
Discharge Follow Up Questionnaire | prior to surgery, up to 2-6 weeks after discharge from the hospital
  Measured with "Yes" or "No", patients were asked if they completed Enhanced Recovery After Surgery (ERAS) protocols and prior to surgery.
Collection of Discharge Disposition | from admission to discharge, up to 20 days
  • Collection of discharge disposition following hospital discharge
Compliance During Hospitalization | from admission to discharge, up to 20 days
  * Compliance with OR checklist
  * Compliance with inpatient ERAS wound care regimen
Patient Reported Outcomes EQ-5D | prior to surgery, up to 6 months after surgery
  Using the EQ-5D, data is collected on a scale of 1 to 3 with 1 being no problem, 2 being moderate problem and 3 being severe problem.
Patient Reported Outcomes EQ-5D (health scale) | prior to surgery, up to 6 months after surgery
  Using the EQ-5D, data is collected health scale for today. On a scale 0 to 100 with 100 being the best health and 0 means the worst health.
Patient Reported Outcomes Oswestry Low Back Pain Disability Questionnaire | prior to surgery, up to 6 months after surgery
  Using the oswestry low back pain disability index (ODI) scale, patients' responses are calculated on a scale of 0 to 100 with 0 being no pain and 100 being the worst pain.
Patient Reported Outcomes Neck Disability Index | prior to surgery, up to 6 months after surgery
  Using the neck pain disability index (NDI) scale, patients' responses are calculated on a scale of 0 to 100 with 0 being no pain and 100 being the worst pain.
Patient Reported Outcomes Neurosurgery Patient Satisfaction | prior to surgery, up to 6 months after surgery
  Using the Neurosurgery Patient Satisfaction Outcome questionnaire, patients' satisfaction are recorded with "Yes" or "No" to questions.
Collection of Working Status | prior to surgery, up to 6 months after surgery
  Collection of patient working status including:
  * currently working
  * retired
  * disabled
  * not working due to a reason other than the condition being treated
Consults | Prior to surgery
  • Rate of provider recommendation for additional consultations
Enhanced Recovery at Penn (ERAP) Text Messaging Program - Patient Enrollment | Up to 3 months after surgery
  • Patient enrollment in service
Enhanced Recovery at Penn (ERAP) Text Messaging Program - Compliance | Up to 3 months after surgery
  • ERAP compliance with carbohydrate loading and surgical site preparation
Enhanced Recovery at Penn (ERAP) Text Messaging Program - Pain Score | Up to 3 months after surgery
  • Pain scores (1 to 10 with 1 being no pain and 10 being worst) at 1, 2, and 3 weeks and at 1, 2, and 3 months postop
Enhanced Recovery at Penn (ERAP) Text Messaging Program - Pain Medication | Up to 3 months after surgery
  * Pain medication use at 1, 2, and 3 weeks and at 1, 2, and 3 months postop
  * Patient engagement and likelihood to recommend text messaging service
Enhanced Recovery at Penn (ERAP) Text Messaging Program - Engagement | Up to 3 months after surgery
  • Patient engagement and likelihood to recommend text messaging service

CONTACTS AND LOCATIONS:
Overall Officials: Zarina Ali, MD, Principal Investigator — University of Pennsylvania; Neil Malhotra, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States